CLINICAL TRIAL: NCT04054557
Title: Utilization of Patient Reported Outcomes Generated by Electronic Medical Record and Smart Pill Bottles With Follow up Telehealth Encounters to Improve Adherence to Adjuvant Endocrine Therapy in Breast Cancer Patients
Brief Title: Patient Reported Outcomes, Smart Pill Bottle and Teleheath for Endocrine Therapy Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18D.003; JT 11620 (Other: JeffTrial Number)
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Stage 0 Breast Cancer AJCC v6 and v7; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage III Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms | interventions — Telemedicine; Practice Guidelines as Topic; Standard of Care; Behavior Therapy; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (Standard of Care office Visits) (Active Comparator): Participants receive standard of care office visits approximately every 3 months (± 2 weeks) for one year.
  Interventions: Other: Best Practice; Other: Questionnaire Administration; Other: Quality-of-Life Assessment
- Arm II (Standard of Care Office Visits, survey, telehealth) (Experimental): Patients receive standard of care as in Arm I and 4 automated electronic surveys every 3 weeks (+/- 1 weeks) for a total of 18 electronic surveys over one year. Patients who report severe or very severe side effects, or stopping or are thinking about stopping their ET will have a follow up encounter with a research coordinator.
  Interventions: Other: Telemedicine; Other: Best Practice; Other: Questionnaire Administration; Other: Quality-of-Life Assessment; Other: Survey Administration
- Arm III (Smart Pill Bottle, messaging) (Experimental): Patients receive a wireless smart pill bottle that performs daily time-specific reminders to open the pill bottle and take the medication. Additional messages are triggered by the pill bottle when non-adherence is indicated (lack of bottle opening or no change in remaining pills), as well as when medication is skipped.
  Interventions: Other: Questionnaire Administration; Other: Quality-of-Life Assessment; Behavioral: Behavioral Intervention; Other: Educational Intervention

INTERVENTIONS:
Other: Telemedicine — Participate in virtual visits with oncologist
  Other Names: Telehealth, telemedicine
  Arms: Arm II (Standard of Care Office Visits, survey, telehealth)
Other: Best Practice — Receive 4 in-office visits with oncologist
  Other Names: best practice, standard of care, standard therapy
  Arms: Arm I (Standard of Care office Visits); Arm II (Standard of Care Office Visits, survey, telehealth)
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Complete electronic survey
  Arms: Arm II (Standard of Care Office Visits, survey, telehealth)
Behavioral: Behavioral Intervention — Use smart pill bottle
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Treatment; Behavioral Interventions
  Arms: Arm III (Smart Pill Bottle, messaging)
Other: Educational Intervention — Receives time-specific reminders and messages
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention; Educational
  Arms: Arm III (Smart Pill Bottle, messaging)

SUMMARY:
This phase II trial studies how well telehealth works in improving adherence to endocrine (anti-estrogen) therapy in participants with estrogen receptor and/or progesterone receptor positive (hormone receptor positive) stage 0-III breast cancer who have underwent surgery. Telehealth is an approach to care that uses digital information and communication tools to manage health and well-being. Participants interact with their health care providers via a video chat on a computer or smart phone. Telehealth may help identify the effects of treatment on participants with breast cancer who have underwent surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate if the utilization of automated patient reported outcomes and follow up Telehealth can improve patient adherence with adjuvant endocrine therapy during the first 12 months of study participation.

II. To evaluate if the utilization of Smart Pill Bottles and follow-up Telehealth encounters can improve patient adherence with adjuvant endocrine therapy during the first 12 months of study participation.

SECONDARY OBJECTIVES:

I. To evaluate if the utilization of automated patient reported outcome and follow-up Telehealth encounters can improve quality of life and decrease side effects while taking adjuvant endocrine therapy.

OUTLINE: Participants are randomized to 1 of 3 arms.

ARM I: Patients receive standard of care office visits approximately every 3 months for one year.

ARM II: Patients receive standard of care as in Arm I and 4 automated electronic surveys every 3 weeks (+/- 1 weeks) for a total of 18 electronic surveys over one year. Patients who report severe or very severe side effects, or stopping or are thinking about stopping their endocrine therapy (ET) will have a follow up encounter with a research coordinator.

ARM III: Patients receive a wireless smart pill bottle that performs daily time-specific reminders to open the pill bottle and take the medication. Additional messages are triggered by the pill bottle when non-adherence is indicated (lack of bottle opening or no change in remaining pills), as well as when medication is skipped.

ELIGIBILITY:
Inclusion Criteria:

* • Signed informed consent obtained prior to any study specific assessments and procedures

  * Eastern Cooperative Oncology Group (ECOG) performance status 0-2
  * Women or men diagnosed with stage 0-III hormone receptor positive (estrogen receptor positive [ER] and /or progesterone receptor [PR] positive) breast cancer

    * Staging for eligibility should utilize the most recent American Joint Committee on Cancer (AJCC) breast cancer staging version
  * Patients (Pts) must have undergone breast surgery for their diagnosis of breast cancer
  * Adjuvant endocrine therapy has been prescribed by their treating physician

    * Patients may receive concurrent adjuvant radiation therapy plus endocrine therapy in the post-operative setting
  * Have a cell phone with text messaging ability
  * Have access to a computer, tablet, or smart phone to complete electronic surveys
  * Patient must be willing to setup an online Jefferson MyChart account
  * Patients who have been on endocrine therapy for more than 4 years

Exclusion Criteria:

* Pts with stage IV metastatic breast cancer
* Patients unable to participate in patient portal communication (e.g. do not have either a smart phone, laptop, access to a computer and/ or access to a device with a webcam)
* Pts who are non-English speaking and English illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Adherence to endocrine therapy (ET) | Up to one year
  ET is defined as the proportion of patients with filled prescriptions to cover >= 80% of their ET doses for the year and pill diaries documenting receipt of >= 80% of prescribed doses of ET for the year. ET medication adherence will be evaluated by pill diary collected at each quarterly clinic visit.

SECONDARY OUTCOMES:
Quality of life assessment | 1 year post intervention
  Patients will fill out the Functional Assessment of cancer Therapy-Endocrine Subscale (FACT-ES) at initiation of trial, and then at each of the quarterly clinic visits for Arm B and on paper for patients on Arm A. The FACT-ES, has two sections each of which will be evaluated separately. The first section, FACT-G, will be used as a measure of general quality of life. It consists of 27 items, each scored 0 to 4. Scores range from 0 to 108 with higher scores indicating worse quality of life.
ET side effects | Up to one year
  Patients will fill out the Functional Assessment of cancer Therapy-Endocrine Subscale (FACT-ES) at initiation of trial, and then at each of the quarterly clinic visits. The FACT-ES, has two sections each of which will be evaluated separately. The second section of the FACT-ES will be used as a measure of specific side effects of endocrine therapy. It consists of 19 items scored 0 to 4 with scores ranging from 0 to 76. A higher score indicates worse side effects. The FACT-ES has established validity and reliability in breast cancer patients.
Satisfaction with cancer care | At 12 months
  This will be evaluated using a modified version of the Patient Satisfaction With Cancer Care Scale (PSCCS). The modified scale contains 14 items, each rated on a 5-point scale ranging from strongly agree (5) to strongly disagree (1). Scores range from 14 to 70 with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Maysa Abu-Khaaf, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (5):
- United States (5):
  - Jefferson Health - South Jersey, Washington Township, New Jersey
  - Thomas Jefefrson University, Philadelphia, Pennsylvania
  - Methodist Hospital, Philadelphia, Pennsylvania
  - Jefferson Health - Northeast, Torresdale, Pennsylvania
  - Jefferson Health - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania

IPD SHARING:
Plan to Share IPD: No